CLINICAL TRIAL: NCT04906304
Title: Comparison of Safety and Efficacy of de Novo Everolimus Plus Low Dose of Cyclosporine With Standard Dose of Cyclosporine Plus Cellcept on CMV and BK Virus Infections Prevention in Renal Transplant Patients
Brief Title: Comparison of Safety and Efficacy of de Novo Everolimus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, assistant Professor of SBMU, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNRC940401/18
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Everolimus; lactitol; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evrolimus (Experimental): The treatment regimen in everolimus group was 0.75 mg/bid everolimus with everolimus C0 3-8 ng/mL plus Sandimmun (Neoral) low dose pluse cellcept
  Interventions: Drug: Everolimus Pill; Drug: Sandimmun (Neoral) dose plus cellcept
- Control (Active Comparator): 0.75 mg/bid everolimus with everolimus C0 3-8 ng/mL plus Sandimmun (Neoral)standard dose plus cellcept
  Interventions: Drug: Everolimus Pill; Drug: Sandimmun (Neoral) dose plus cellcept

INTERVENTIONS:
Drug: Everolimus Pill — standard dose versus low dose Sandimun
  Other Names: Novartis
Drug: Sandimmun (Neoral) dose plus cellcept — Sandimmun (Neoral) dose plus cellcept

SUMMARY:
Nowadays, de novo everolimus regimen in renal transplant patients is considered for reduction of cyclosporine dose and it is mentioned that this regimen not only has similar safety and efficacy, but also could prevent Cytomegalovirus (CMV )infections. So, the aim of this study was comparison of safety and efficacy of de novo everolimus plus low dose of cyclosporine with standard dose of cyclosporine plus cellcept on CMV virus infections prevention in renal transplant patients.

DETAILED DESCRIPTION:
This randomized clinical trial was conducted in Shahid Labbafi nejad hospital. 35 renal transplanted patients enter the study and randomized to one of two groups: everolimus or control (Sandimmun or tacrolimus). However, 34 patients completed study (17 patients in each group). The treatment regimen in everolimus group was 0.75 mg/bid everolimus with everolimus C0 3-8 ng/mL plus Sandimmun (Neoral) low dose and in control group was standard dose of Sandimmun or tacrolimus plus cellcept. All patients gave Antithymocyte Glubolin and prednisolone. In addition, they gave CMV prophylaxis until 3 months. Kidney biopsies were done for raise of creatinine or protocol biopsy at 6 month after transplantation. Demographic, renal disease and transplantation characteristics, CMV and BK virus status, rejection, and routine laboratory tests recorded during study period and compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult Transplanted patients > 18 years

Exclusion Criteria:

* Simultanous Kidney -Pancreas Transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
CMV Infection | 6 months
  CMV PCR quantitative count

CONTACTS AND LOCATIONS:
Overall Officials: SBMU University of Medical Sciences, Study Director — Shahid Beheshti University of Medical Sciences
Locations (1):
- Nooshin Dalili, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No